CLINICAL TRIAL: NCT03690193
Title: Alzheimer's Disease Ketogenic Diet Retention and Feasibility Trial
Brief Title: Feasibility and Efficacy of the Ketogenic Diet in Alzheimer's Disease
Acronym: KDRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Debra K. Sullivan, PhD, RD, Debra K Sullivan, PhD, RD, Chair and Endowed Professor of Clinical Nutrition, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13796
Record Dates: First submitted 2018-08-01; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Alzheimer Disease
Keywords: Ketogenic Diet; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet Arm (Experimental): All participants will be assigned to the 3-month ketogenic diet intervention. Study partners will be instructed to assist participants in adherence to a 1:1 ketogenic diet (approximately 70% fat, <10% carbohydrate, and 20% protein). Participants will be provided medium chain triglyceride oil with a target intake of 1-2 tablespoons per day and micronutrient supplements consisting of multivitamin, vitamin D, calcium, and phosphorus. After the 3-month ketogenic diet, participants will complete a 1-month washout period in which they halt adherence to the ketogenic diet and resume their normal diet.
  Interventions: Behavioral: Ketogenic Diet

INTERVENTIONS:
Behavioral: Ketogenic Diet — All participants will be assigned to the 3-month 1:1 ketogenic diet intervention (approximately 70% fat, <10% carbohydrate, and 20% protein).

SUMMARY:
The purpose of the KDRAFT study is to assess the feasibility and preliminary cognitive efficacy of a ketogenic diet therapy in patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease (CDR 0.5, 1, & 2)
* Active study partner
* BMI > 21
* English speaking

Exclusion Criteria:

* BMI < 21
* Consume greater than 14 drinks of alcohol per week
* Insulin Dependent Diabetes Mellitus
* Diagnosis of active cancer
* Myocardial infarction or symptoms of coronary artery disease (e.g. angina) in last year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-06 (Actual)

PRIMARY OUTCOMES:
Proportion of days positive for urinary ketone production | Daily for 90 days (the length of the diet intervention)
  Participants will measure and report daily urinary ketone status using Ketostix (Bayer, Germany).
Change in blood ketone levels induced by ketogenic diet | Change from baseline serum beta-hydroxybutyrate levels at month 1, 2, 3 (end of ketogenic diet), and 4 (after 1-month washout).
  Serum beta-hydroxybutyrate levels will be measured at five monthly study visits; baseline prior to diet initiation, three monthly collections during the ketogenic diet intervention, and after the 1-month washout return to a regular diet.

SECONDARY OUTCOMES:
Change in cognitive performance on the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) | Change from baseline global cognitive scores at month 3 (end of ketogenic diet) and change from month 3 global cognitive scores at month 4 (end of 1-month washout).
  Global cognitive performance will be assessed by a psychometrician using the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog). The ADAS-Cog is an Alzheimer's disease specific, multi-domain cognitive assessment scored from 0-70 points with higher scores indicating poorer cognitive performance.
Change in cognitive performance on the Mini-Mental State Exam (MMSE) | Change from baseline global cognitive scores at month 3 (end of ketogenic diet) and change from month 3 global cognitive scores at month 4 (end of 1-month washout).
  Global cognitive performance will be assessed by a psychometrician using the Mini-Mental State Exam (MMSE). The MMSE is a brief cognitive questionnaire with a maximum score of 30 points where higher scores indicate better cognitive performance.
Dietary intake characterization prior to and after ketogenic diet initiation | Dietary intake will be collected at Baseline, Month 1, Month 2, Month 3
  Changes in food and nutrient intake will be assessed by monthly 3-day food records completed by participant study partners.

REFERENCES:
- [Derived] Taylor MK, Swerdlow RH, Burns JM, Sullivan DK. An Experimental Ketogenic Diet for Alzheimer Disease Was Nutritionally Dense and Rich in Vegetables and Avocado. Curr Dev Nutr. 2019 Feb 20;3(4):nzz003. doi: 10.1093/cdn/nzz003. eCollection 2019 Apr. PMID 30931426